CLINICAL TRIAL: NCT04598581
Title: Low Dose Radiation Therapy for Severe-Acute-Respiratory-Syndrome-Coronavirus-2 (SARS-CoV-2)
Brief Title: Low Dose Radiation Therapy for Severe-Acute-Respiratory-Syndrome-Coronavirus-2 (SARS-CoV-2), COVID-19
Acronym: COVID-RT-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-02047qu20Papachristofilou
Record Dates: First submitted 2020-10-20; First posted 2020-10-22 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Severe-Acute-Respiratory-Syndrome-Coronavirus-2 (SARS-CoV-2)
Keywords: Low dose radiation therapy (LD-RT)
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Information on group allocation will not be disclosed to either the patient or the ICU-staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Dose Radiation Therapy (LD-RT) (Active Comparator)
  Interventions: Radiation: Low Dose Radiation Therapy (LD-RT)
- Sham irradiation (Sham Comparator)
  Interventions: Other: Sham irradiation

INTERVENTIONS:
Radiation: Low Dose Radiation Therapy (LD-RT) — Low Dose Radiation Therapy (LD-RT) of both lungs with 1 Gray
  Arms: Low Dose Radiation Therapy (LD-RT)
Other: Sham irradiation — Sham irradiation
  Arms: Sham irradiation

SUMMARY:
This study is to analyse the efficacy of LD-RT for treatment of Severe-Acute-Respiratory-Syndrome-Coronavirus-2 (SARS-CoV-2).

DETAILED DESCRIPTION:
Management of patients with SARS-CoV-2 presents a great challenge in the ongoing pandemic. The inflammatory reaction, evident in the later stages of the disease, is linked with high mortality rates. Pharmaceutical interventions at this stage often do not achieve the desired effects. Low Dose Radiation Therapy (LD-RT) has been utilized for treatment of inflammatory conditions because of its immunomodulatory effects. Thus, LD-RT may be an option in SARS-CoV-2 based on pre-clinical models and early clinical data. This study is to analyse the efficacy of LD-RT for treatment of Severe-Acute-Respiratory-Syndrome-Coronavirus-2 (SARS-CoV-2).

ELIGIBILITY:
Inclusion Criteria:

* Age of male patients >40 years
* Age of female patients >50 years
* Patients with SARS-CoV-2 requiring mechanical ventilation
* Informed consent obtained by the legal representative of the patient

Exclusion Criteria:

* Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Ventilator free days (VFD) | at day 15 after LD-RT
  Ventilator free days (VFD)

SECONDARY OUTCOMES:
Change in pulmonary function, measured as relative change (%) from baseline in oxygenation index (PaO2 / FiO2) | at day 5, 10, 15, 28 after LD-RT
  Change in pulmonary function, measured as relative change (%) from baseline in oxygenation index (PaO2 / FiO2)
Overall mortality | at day 15 and 28 after LD-RT
  Overall mortality
Change in levels of ferritin (ng/ml) | up to day 15 after LD-RT
  Change in levels of ferritin (ng/ml)
Change in levels of c-reactive protein (mg/l) | up to day 15 after LD-RT
  Change in levels of c-reactive protein (mg/l)
Change in levels of white blood cell counts (number of white blood cells per volume of blood) | up to day 15 after LD-RT
  Change in levels of white blood cell counts (number of white blood cells per volume of blood)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Papachristofilou, Dr. med., Principal Investigator — Department of Radiooncology, University Hospital Basel
Locations (1):
- Department of Radiooncology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Papachristofilou A, Finazzi T, Blum A, Zehnder T, Zellweger N, Lustenberger J, Bauer T, Dott C, Avcu Y, Kohler G, Zimmermann F, Pargger H, Siegemund M. Low-Dose Radiation Therapy for Severe COVID-19 Pneumonia: A Randomized Double-Blind Study. Int J Radiat Oncol Biol Phys. 2021 Aug 1;110(5):1274-1282. doi: 10.1016/j.ijrobp.2021.02.054. Epub 2021 Mar 5. PMID 33677049